CLINICAL TRIAL: NCT05133128
Title: An Experimental Medicine, Low Grade Interventional, Clinical Study to Compare Peripheral Immune System From Subjects Without Cancer Diagnosis and Patients With Advanced Solid Tumours
Brief Title: An Experimental Medicine Clinical Study to Compare Peripheral Immune System From Subjects Without Cancer Diagnosis and Patients With Solid Tumours.
Acronym: IMMUNOPBMC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of promotor
Sponsor: Servier (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A01796-35
Record Dates: First submitted 2021-11-15; First posted 2021-11-24 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Immune System
Keywords: PBMC; cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PATIENTS with cancer and HEALTHY VOLUNTEERS (Other): * Cohort 1: Patients with Non-Small Cell Lung cancer (25 patients)
  * Cohort 2: Patients with Colorectal cancer (25 patients)
  * Cohort 3: Patients with Pancreatic cancer (25 patients)
  * Cohort 4: Patients with Liver cancer (25 patients)
  * Cohort 5: Patients with Gastric cancer/cholangiocarcinoma (25 patients)
  * Cohort 6: Healthy volunteers (25 subjects)
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — blood samples

SUMMARY:
The aim of the study is to gain knowledge concerning expression of immune markers on immune cell subpopulation of PBMCs from subjects without cancer diagnosis and cancer patients. Few studies have addressed the question of the difference of peripheric immune cells between these two populations without a specific focus on an immune cell population or an indication, and with a multiparametic approach. The present study will combine phenotypic (using cell population markers and immune checkpoints) and functional analyses toallow to better interpret non-clinical results obtained with either subjects without cancer or cancer patient material and provide rationale to use material from subjects without cancer diagnosis for functional tests. It would also argument a go to healthy volunteer's clinical trials for assessing peripheral pharmacodynamic (PD), receptor occupancy (RO) and safety (Cytokine release syndrome, CRS), in the context of early drug development in immuno-oncology. Finally, generated data will be used to feed quantitative system pharmacology (QSP) models to increase their robustness and better predict drug pharmacology in humans.

ELIGIBILITY:
• INCLUSION CRITERIA FOR ALL PARTICIPANTS (PATIENTS WITH CANCER AND HEALTHY VOLUNTEERS)

1. The participating subjects are able to provide signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
2. Men and women must be of 45 to 70 years of age on the day the consent is signed. Non-cancer subjects should be age matched by +/- 5 years with the cancer patient population.
3. Subject must have a Negative HIV
4. Adequate hematological parameters as assessed by laboratory tests within 21 days for cancer patients and 96 hours for healthy volunteers prior to the day of blood withdrawal:

   1. Absolute Neutrophil Count (ANC) ≥1500/µL
   2. Platelet count ≥100 000/µL, criteria must be met without transfusion and thrombopoietin for at least two weeks prior to the day of blood withdrawal
   3. Hemoglobin ≥9g/dL, criteria must be met without transfusion and erythropoietin for at least two weeks prior to the day of blood withdrawal
5. Physical ability to tolerate a 60 ml-blood sampling.
6. Subjects affiliated to a social security regimen or beneficiary of the same according to local requirements

   • INCLUSION CRITERIA FOR CANCER PATIENTS ONLY
7. Patients currently off treatment with histologically or cytologically confirmed following diagnosis:

   * Cohort 1: Unresectable, locally advanced or metastatic Non-Small Cell Lung cancer after at least 1 or 2 standard treatment lines (including 1 line with Immune Checkpoint Inhibitor) and being scheduled for a new anti-cancer treatment after progression
   * Cohort 2: Unresectable, locally advanced or metastatic Colorectal cancer after at least 2 treatment lines
   * Cohort 3: Unresectable, locally advanced or metastatic Pancreatic cancer after at least 1 or 2 treatment lines
   * Cohort 4: Unresectable, locally advanced or metastatic Liver cancer before or after at least 1 treatment line
   * Cohort 5: Unresectable, locally advanced or metastatic Gastric cancer after at least 1 treatment line Unresectable, locally advanced or metastatic Cholangiocarcinoma before or after at least 1 treatment line

     * NON-INCLUSION CRITERIA FOR ALL PARTICIPANTS (PATIENTS WITH CANCER AND HEALTHY VOLUNTEERS)
8. Pregnant women
9. Subjects with an active autoimmune disease that is currently requiring systemic anti-inflammatory treatment such as disease-modifying anti-rheumatic drugs [DMARDs], steroids, or immunosuppressants), except vitiligo, alopecia areata, asthma/atopy and psoriasis treated and controlled by topical therapies. Patients with auto-immune endocrinopathies that are well treated by replacement hormones therapies (e.g. thyroxine, insulin, physiological steroids for adrenal or pituitary) are allowed. Patients with a history of immune related adverse events (irAEs) from a previous line of treatment must have resolved their irAEs to a grade ≤1 and have stopped any immunosuppressive/steroid therapy
10. Subjects with any serious/active/uncontrolled infection, any infection requiring parenteral antibiotics, or unexplained fever >38ºC within 2 weeks prior to blood withdrawal.
11. Subjects who have had a laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) test within 60 days prior to blood withdrawal.
12. Patients seropositive for and with evidence of active viral infection with hepatitis B virus (HBV). Patients who are hepatitis B surface antigen (HBsAg) negative and HBV viral DNA negative are eligible.

    1. Patients who had HBV but have received an antiviral treatment and show non-detectable viral DNA for 6 months are eligible.
    2. Patients who are seropositive because of HBV vaccine are eligible. Note: a quantitative PCR test result of < 10 IU/mL is equivalent to being undetected (negative). Subject with no available results for hepatitis B virus (HBV) are eligible.
13. Patients seropositive for and with active viral infection with hepatitis C virus (HCV). Patients who had HCV but have received an antiviral treatment and show no detectable HCV viral DNA for 6 months are eligible.

    Note: a quantitative PCR test result of < 10 IU/mL is equivalent to being undetected (negative). Subject with no available results for hepatitis C virus (HCV) are eligible.
14. Subjects who have received prior systemic anticancer therapy, definitive radiotherapy (palliative radiation therapy is allowed), or other investigational agents or device within 14 days prior to the day of blood withdrawal (or 5 half-lives of the therapeutic agents whatever the shortest). Patients who are in the screening period of an investigational study may participate if they are currently off-treatment. Patients who have entered the follow-up period of an investigational study may participate if it has been 2 weeks after the last dose of the previous investigational agent.
15. Subjects who have received approved or investigational immunomodulators (targeting any immune cell types, such as anti-CTLA-4, anti-PD-L1, any immunomodulatory in a clinical trial) in the past 6 months (except for the NSCLC cohort).
16. Subjects who have not recovered from the effects of a major surgery.
17. Subject under guardianship, curatorship or safeguard of justice
18. Subjects who have received a vaccine within 60 days prior to blood withdrawal.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Standard differential blood count | 1 day
  flow cytometry analysis

CONTACTS AND LOCATIONS:
Overall Officials: François GHIRINGHELLI, PU-PH, Principal Investigator — Centre Georges François Leclerc
Locations (2):
- France (2):
  - Centre Georges Francois Leclerc, Dijon
  - CIC du CHU, Dijon